CLINICAL TRIAL: NCT02868489
Title: Effect of Bacillus Coagulans and Galactomannans on Obese Patients Undergoing Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Keith Scharf, DO, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5160281
Record Dates: First submitted 2016-07-28; First posted 2016-08-16 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Quality of Life
Keywords: Microbiota
MeSH Terms: conditions — Obesity | interventions — galactomannan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprietary Blend - LactoWise® (Experimental): After being randomized into two groups, the assigned experimental group, prior to surgery and after consenting, will be asked to complete the Gastrointestinal Quality of Life Index. In addition the experimental group will be given their supply of LactoWise®. They will be required to take 1 capsule per day (300 mg of bacillus coagulans and galactomannans at 4.5 billion live cells) at breakfast consistently for 3 months. There will be three follow up visits (Week-2, Week-6 and Month-3) where participants will be asked to complete the gastrointestinal quality of life index.
  Interventions: Dietary Supplement: LactoWise®
- Control (Placebo Comparator): For the control group, prior to surgery and after consenting to enroll in the study participants will also be asked to complete the Gastrointestinal Quality of Life Index. Participants of the control group will be administered their supply of a matching placebo. They will be required to take 1 capsule per day at breakfast consistently for 3 months. There will be three follow up visits (Week-2, Week-6 and Month-3) where participants will be asked to complete the gastrointestinal quality of life index.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LactoWise® — blend of bacillus coagulans and galactomannans
  Other Names: blend of bacillus coagulans and galactomannans
  Arms: Proprietary Blend - LactoWise®
Other: Placebo — Placebo to be selected is calcium carbonate (since participant routine standard of care already includes intake of calcium citrate)
  Arms: Control

SUMMARY:
The purpose of the study is to determine the effect of bacillus coagulans and galactomannans (LactoWise®) administration on obese patients undergoing sleeve gastrectomy by observing standard protocol measurements in patients following sleeve gastrectomy: laboratory measurements, ideal body weight, and percent estimated weight loss, in addition incorporating the Gastrointestinal Quality of Life Index (GIQLI)

DETAILED DESCRIPTION:
Loma Linda University's School of Allied Health Professions in collaboration with the Metabolic and Bariatric Surgery Department under the Surgery Division is conducting research to evaluate the influence of LactoWise® (a proprietary blend of probiotic and prebiotic - bacillus coagulans/galactomannans, respectively) on the normal microbiota of obese patients post bariatric sleeve gastrectomy. Pre-surgery, participants will be required to sign a consent form and to complete the Gastro-Intestinal Quality of Life Index (GIQLI). A total of 60 bariatric sleeve patients will be recruited for this investigation. Post-surgery participants will be randomized into two groups, one will receive LactoWise® and one be the control (placebo). The LactoWise® blend has 300 mg of the bacillus coagulans and galactomannans and contains around 4.5 billion live cells. Daily intake of capsules coupled with bariatric sleeve standard of care will be conducted for the duration of 3 months, which is the anticipated clinical timeline. Participants will also be asked to complete the quality of life questionnaire at each of the following follow-ups post-surgery: 2nd week, 6th week, and 3rd month.

Outcome measures will be the standard protocol for bariatric sleeve patients at the Metabolic and Bariatric Surgery Department which will include weight measurements, blood work. In addition to the standard of care procedures a research procedure to be added is the GIQLI. Pre and post clinical consults, administration of probiotic/prebiotic formulae, and follow-ups will be conducted at the Faculty Medical Offices - General Surgery - Bariatric Clinic at Loma Linda University Health.

ELIGIBILITY:
Inclusion Criteria:

* Patient of bariatric sleeve surgery
* Ages 18-70
* Consent to complete GIQOL questionnaire
* Commit to consistent use of LactoWise® or placebo assigned for study period

Exclusion Criteria:

* None sleeve bariatric surgery patient
* Have compromised immunity or poorly controlled systems
* Presence of any concurrent active infection
* Physically disabled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Changes in weight percent EWL | Baseline - 3 months
  Changes in weight expressed will be based off of the percent excess body weight loss (percentage EBWL) which is the weight loss relative to ideal weight expressed as a percentage. For the calculation of percentage EBWL the ideal body weight will be based off of BMI 25. BMI will be measured in kg/m^2. Studies have shown that changes in the physical structure or manipulation of the gastrointestinal system may influence normal microbiota which can be characterized by changes in metabolism which in turn will be tested by changes in weight

CONTACTS AND LOCATIONS:
Overall Officials: Keith Scharf, DO FACS, Principal Investigator — Loma Linda University Health
Locations (1):
- Faculty of Medical Offices - LLU, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodard GA, Encarnacion B, Downey JR, Peraza J, Chong K, Hernandez-Boussard T, Morton JM. Probiotics improve outcomes after Roux-en-Y gastric bypass surgery: a prospective randomized trial. J Gastrointest Surg. 2009 Jul;13(7):1198-204. doi: 10.1007/s11605-009-0891-x. Epub 2009 Apr 18. PMID 19381735